CLINICAL TRIAL: NCT06063876
Title: Progression and Resolution of Experimental Peri-implant Mucositis on Now Healthy Implant Sites That Were Previously Treated With or Without Implantoplasty: A Controlled Clinical Trial
Brief Title: Experimental Peri-implant Mucositis on Implant Sites That Were Previously Treated With or Without Implantoplasty
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Andrea Ravida, Assistant professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY22060181
Record Dates: First submitted 2023-09-06; First posted 2023-10-03 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis
Keywords: Implantoplasty; Marginal bone level; Probing depth; Bleeding on probing
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implants with history of peri-implantitis (Experimental): Implant(s) treated previously for peri-implantitis with or without exposed polished surface, no PD > 4 mm and < 50% bone loss.
  Interventions: Procedure: Induction of experimental peri-implant mucositis; Procedure: Resolution of experimental peri-implant mucositis

INTERVENTIONS:
Procedure: Induction of experimental peri-implant mucositis — Patients will refrain from oral hygiene measures at the implant sites for 3 weeks to induce peri-implant mucositis, by using a stent in the included implant during oral hygiene.
Procedure: Resolution of experimental peri-implant mucositis — Patients will reinstitute oral hygiene measures, receive an oral prophylaxis and oral hygiene instructions and will be evaluated during 3 weeks.

SUMMARY:
This controlled clinical trial will assess clinically, immunologically, and microbiologically the healing of experimental peri-implant mucositis (PIM) lesions in implants treated previously with implantoplasty (IP) compared to those treated without IP.

DETAILED DESCRIPTION:
The present parallel controlled clinical trial is designed as a 21-day experimental peri-implant mucositis, followed by a period of resolution of 21 days in healthy implants that were previously treated for peri-implantitis with and without implantoplasty.

A total of 8 appointments over the course of about 42 days will be necessary. These appointments will take place in the Department of Periodontics & Preventive Dentistry and are described as follows:

Screening Appointment (14 days prior to Day 0): During this visit, informed consent will be obtained from each subject and inclusion criteria for participation in the study will be reviewed. Participants will undergo the following activities:

* Review of medical, dental history and medications
* Periodontal chart
* Intraoral photographs
* Periapical radiograph of the dental implant that was previously treated with or without implantoplasty to confirm if the implant is in healthy condition with no progressive bone loss
* A digital impression (intraoral scan) of the teeth will be taken for fabrication of a customized stent (a plastic cover). The participant will be instructed to place the stent over the implant whenever performing oral care measures (brushing/flossing/mouthrinse) at home for 21 days. The authors will teach the individuals on how to use this stent and how to brush the teeth/implant(s) during the study. The stent will be provided at the next research visit.
* A professional prophylaxis (dental cleaning) of all tooth and implant surfaces.

V2 - V5 (from day 0 to day 21), the experimentally induced peri-implant mucositis phase, the participant will be wearing the stent over the implant area during their routine oral health care. The following research activities will occur:

* Review any changes to medical or dental history and any new medications
* Intraoral photographs
* Clinical assessment
* Peri-implant crevicular fluid sample collection from the deepest pocket around the implant using paper points.
* Biofilm sample collection using sterile curettes (titanium or plastic) at the same sites.

At V5 (day 21), the participants will receive a dental cleaning, polishing, and review of their oral hygiene home care techniques. Then, they will be asked to reinstitute their oral hygiene home care procedures.

At V6 - V8 (from day 28 to day 42), the resolution of induced peri-implant mucositis phase, the following research activities will occur:

* Review any changes to medical or dental history and any new medications
* Intraoral photographs
* Clinical assessment
* Peri-implant crevicular fluid sample collection from the deepest pocket around the implant using paper points.
* Biofilm sample collection using sterile curettes (titanium or plastic) at the same sites.

At V8 (day 42), a new periapical radiograph will be acquired. If there is still any evidence of inflammation around the implant, we will continue to monitor/treat the inflammation every 3-4 weeks until it is resolved.

PERI-IMPLANT CREVICULAR FLUID (PICF) SAMPLING AND ANALYSIS:

PICF samples will be collected weekly. The site with the deepest pocket of each implant will be sampled using sterile Periopapers with colored bands (29 mm, ISO 25, taper .02; VDW, Munich, Germany). At each visit following screening (V2-V8), the samples will be taken from the same site. The PICF volume will be measured with a calibrated, electronic gingival fluid measuring device (Periotron 8000, Oraflow, Plainview, NY, USA). Cytokines will be detected using a panel of relevant cytokines using a bead based multiplex immunoassay (Bio-Plex Pro Human Cytokine 27-plex Assay).

SUBMUCOSAL PLAQUE SAMPLING AND DNA EXTRACTION Sterile curettes (titanium or plastic) will be used to collect plaque samples from the deepest pocket around each implant. DNA will be extracted using DNeasy Blood and Tissue Kit (Qiagen). Genomic DNA samples will be profiled with 16S Amplicon Sequencing Service. Microbial composition will be profiled with Centrifuge using bacterial, viral, fungal, and human genome datasets.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years
* In good general health, (at least ASA 2)
* Previously treated implants must have probing depths (PD) ≤ 4 mm
* Previously treated implants must have <50% bone loss around the implant of interest (assessed radiographically)
* Patients must have been treated previously for peri-implantitis with or without IP, with at least 1 thread or 2 mm of implant surface exposed in the oral cavity.
* Have little to no bacteria on the implant(s) of interest (modified Plaque Index of <1) by Day 0
* Have healthy gums that do not bleed around the implant(s) of choice (modified Gingival index <1) by Day 0
* Have evidence of stable bone levels around the treated implant for > 6 months

Exclusion Criteria:

* Active infectious diseases of any kind.
* Medical conditions which require premedication prior to dental treatments/visits.
* Pregnant women or planning to become pregnant (self-reported).
* Patients with congenital or metabolic bone disorders (ie. osteoporosis, vitamin D deficiency, parathyroid disease, etc.)
* Current heavy smokers: Subjects who have smoked more than 1 pack/day within 6 months of study onset (self-reported)
* Subjects with co-morbid conditions (i.e., uncontrolled diabetes, cardiovascular disease, impaired kidney function, heart murmur, rheumatic fever, bleeding disorder, hepatitis, tuberculosis, HIV) that would affect the study outcome or interpretation of study results will be excluded.
* Concomitant medications: Subjects on significant concomitant drug therapy for systemic conditions (i.e., Chronic anti-inflammatory medication, antibiotics, anticoagulants, any medication initiated <3 months prior to the screening visit) will not be included in the study. Occasional short-term use (7-14 days) of analgesics or common cold medication is permitted. Such use of these medications will be reviewed and recorded by the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the modified Gingival Index (mGI) between 21 and 42 days | At 21 and 42 days
  The mGI will be assessed according to the following criteria:
  Score 0 - No bleeding on probing; Score 1 - Bleeding dot; Score 2 - Continuous line of blood that fills the sulcus; Score 3 - Profuse bleeding and/or hemorrhage drip.
  Changes in the scores between day 21 and day 42 will be determined, being 0 minimum and 3 maximum. The mGI will be assessed weekly.

SECONDARY OUTCOMES:
modified Plaque Index (mPI) | Up to 42 days
  The mPI will be assessed according to the following criteria:
  Score 0 - No visible plaque; Score 1 - Plaque only recognized by running a probe across the marginal surface; Score 2 - Plaque can be seen by the naked eye; Score 3 - Abundance of soft matter
  The mPI will be assessed weekly, being 0 minimum and 3 maximum.
Changes in probing depth (PD) | Up to 42 days
  PD will be accessed weekly. Increase in PD must exceed a threshold of 0.8mm to be considered progression of the disease.
Marginal bone loss (MBL) | From baseline to 42 days
  Measured by overlaying the baseline and final radiographs and measuring the change in marginal bone levels. Progression will have to exceed a threshold of 0.5mm to be considered.
Peri-implant crevicular fluid (PICF) immunologic profile | Up to 42 days
  PICF will be collected from the same sites weekly with the aid of paper strips. Cytokines will be detected using a panel of relevant cytokines using a bead based multiplex immunoassay to determine the immunological profile of the lesions during induction and resolution of peri-implant mucositis.
Microbiological profile of the biofilm analysis | Up to 42 days
  Plaque samples will be collected weekly and qualitative/quantitatively evaluated by 16S rRNA sequencing for composition profiling during the induction and resolution of peri-implant mucositis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ravida, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Dental Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No